CLINICAL TRIAL: NCT04295200
Title: Changes in Muscle Activity, Squat, and Gait Kinematics After Dry Needling Treatment of the Low Back: A Pilot Study
Brief Title: Muscle Activity and Kinematic Changes With Dry Needling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Principal Investigator, April Brown, Doctor of Physical Therapy, Clinical Instructor, Louisiana State University Health Sciences Center Shreveport
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00001301
Record Dates: First submitted 2020-02-22; First posted 2020-03-04 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Healthy
Keywords: lumbar multifidi; dry needling; electromyography; kinematic
MeSH Terms: interventions — Dry Needling; Electric Stimulation

STUDY DESIGN:
Intervention Model Description: single group pre-test/post-test study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dry needling with electrical stimulation (Experimental): Use of dry needles (this is the generic name for sterile, solid filament needles) are inserted into the lumbar multifidi. Intramuscular electrical stimulation will then be applied by attaching a six-lead electrical stimulation unit to the needles. Electrical stimulation will be applied through the needles at the participant's desired frequency (between 4-6 Hz) and for up to 10 minutes total.
  Interventions: Other: Dry needling with electrical stimulation

INTERVENTIONS:
Other: Dry needling with electrical stimulation — Paravertebral dry needling to L3, 4, 5 multifidi. Electrical stimulation will be applied through the needles for up to 10 minutes total or to the participant's tolerance.

SUMMARY:
This study assesses the effects of dry needling with electrical stimulation to the low back on muscle activity and changes in movement. The investigators hypothesize that dry needling and electrical stimulation will elicit changes in muscle activity as well as changes in movement.

DETAILED DESCRIPTION:
This study will utilize a Vicon motion capture system in conjunction with a Noraxon wireless surface electromyography system to analyze movements and muscle activity of each participant pre and post needling.

ELIGIBILITY:
Inclusion Criteria:

* English speaking individuals between the ages of 18 and 60 years old
* without current complaint of low back pain
* no history of low back or lower extremity surgery

Exclusion Criteria:

* individuals with current complaint of low back pain,
* lumbar radicular symptoms
* history of low back surgery or lower extremity surgery
* pregnancy or planning to become pregnant,
* currently taking immunosuppressant or anticoagulation use with INR not within therapeutic range
* needle phobia
* osteoporosis will be excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-06-16 (Actual)

PRIMARY OUTCOMES:
Muscle activity changes | pre/ post dry needling treatment. Participants' EMG will be recorded over a series of movements of the lumbar spine, will immediately be dry needled with electrical stimulation for up to 10 minutes, then will be immediately reassessed. Total time 2 hours
  activity measured and quantified from the amplitude (mV) of the surface EMG electrodes
Kinematic changes | Participants kinematics will be recorded over a series of movements of the lumbar spine, will immediately be dry needled with electrical stimulation for up to 10 minutes, then will be immediately reassessed. Total time 2 hours
  Measurement of lumbopelvic angles during range of motion activities

CONTACTS AND LOCATIONS:
Overall Officials: April J Brown, DPT, Principal Investigator — LSU Health Science Center Shreveport
Locations (1):
- LSU Health Science Center, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Association APT. Dry needling in clinical practice:an educational resource paper. Alexandria, VA: American Physical Therapy Association; 2013.
- [Background] Therapy FoSBoP. Dry Neelding Resource Paper (Intramuscular Manual Therapy). 4th ed. Alexandria, VA: Federation of State Boards of Physical Therapy; 2013.
- [Background] Caldwell J. Attorney General Opinion 14-0216. In: Justice2015.
- [Background] Koppenhaver SL, Walker MJ, Su J, McGowen JM, Umlauf L, Harris KD, Ross MD. Changes in lumbar multifidus muscle function and nociceptive sensitivity in low back pain patient responders versus non-responders after dry needling treatment. Man Ther. 2015 Dec;20(6):769-76. doi: 10.1016/j.math.2015.03.003. Epub 2015 Mar 13. PMID 25801100
- [Background] Abbaszadeh-Amirdehi M, Ansari NN, Naghdi S, Olyaei G, Nourbakhsh MR. Neurophysiological and clinical effects of dry needling in patients with upper trapezius myofascial trigger points. J Bodyw Mov Ther. 2017 Jan;21(1):48-52. doi: 10.1016/j.jbmt.2016.04.014. Epub 2016 Apr 14. PMID 28167189
- [Background] Haser C, Stoggl T, Kriner M, Mikoleit J, Wolfahrt B, Scherr J, Halle M, Pfab F. Effect of Dry Needling on Thigh Muscle Strength and Hip Flexion in Elite Soccer Players. Med Sci Sports Exerc. 2017 Feb;49(2):378-383. doi: 10.1249/MSS.0000000000001111. PMID 27685009
- [Background] Dunning J, Butts R, Young I, Mourad F, Galante V, Bliton P, Tanner M, Fernandez-de-Las-Penas C. Periosteal Electrical Dry Needling as an Adjunct to Exercise and Manual Therapy for Knee Osteoarthritis: A Multicenter Randomized Clinical Trial. Clin J Pain. 2018 Dec;34(12):1149-1158. doi: 10.1097/AJP.0000000000000634. PMID 29864043
- [Background] Unverzagt C, Berglund K, Thomas JJ. DRY NEEDLING FOR MYOFASCIAL TRIGGER POINT PAIN: A CLINICAL COMMENTARY. Int J Sports Phys Ther. 2015 Jun;10(3):402-18. PMID 26075156
- [Background] Liu L, Huang QM, Liu QG, Thitham N, Li LH, Ma YT, Zhao JM. Evidence for Dry Needling in the Management of Myofascial Trigger Points Associated With Low Back Pain: A Systematic Review and Meta-Analysis. Arch Phys Med Rehabil. 2018 Jan;99(1):144-152.e2. doi: 10.1016/j.apmr.2017.06.008. Epub 2017 Jul 8. PMID 28690077
- [Background] Jayaseelan DJ, Moats N, Ricardo CR. Rehabilitation of proximal hamstring tendinopathy utilizing eccentric training, lumbopelvic stabilization, and trigger point dry needling: 2 case reports. J Orthop Sports Phys Ther. 2014 Mar;44(3):198-205. doi: 10.2519/jospt.2014.4905. Epub 2013 Nov 21. PMID 24261928
- [Background] Rainey CE. The use of trigger point dry needling and intramuscular electrical stimulation for a subject with chronic low back pain: a case report. Int J Sports Phys Ther. 2013 Apr;8(2):145-61. PMID 23593553
- [Background] Koppenhaver SL, Walker MJ, Rettig C, Davis J, Nelson C, Su J, Fernandez-de-Las-Penas C, Hebert JJ. The association between dry needling-induced twitch response and change in pain and muscle function in patients with low back pain: a quasi-experimental study. Physiotherapy. 2017 Jun;103(2):131-137. doi: 10.1016/j.physio.2016.05.002. Epub 2016 May 20. PMID 27623385
- [Background] Dar G, Hicks GE. The immediate effect of dry needling on multifidus muscles' function in healthy individuals. J Back Musculoskelet Rehabil. 2016 Apr 27;29(2):273-278. doi: 10.3233/BMR-150624. PMID 26406203
- [Background] Ge HY, Fernandez-de-Las-Penas C, Yue SW. Myofascial trigger points: spontaneous electrical activity and its consequences for pain induction and propagation. Chin Med. 2011 Mar 25;6:13. doi: 10.1186/1749-8546-6-13. PMID 21439050
- [Background] Lucas KR, Rich PA, Polus BI. Muscle activation patterns in the scapular positioning muscles during loaded scapular plane elevation: the effects of Latent Myofascial Trigger Points. Clin Biomech (Bristol). 2010 Oct;25(8):765-70. doi: 10.1016/j.clinbiomech.2010.05.006. Epub 2010 Jul 27. PMID 20667633
- [Background] Ge HY, Monterde S, Graven-Nielsen T, Arendt-Nielsen L. Latent myofascial trigger points are associated with an increased intramuscular electromyographic activity during synergistic muscle activation. J Pain. 2014 Feb;15(2):181-7. doi: 10.1016/j.jpain.2013.10.009. Epub 2013 Nov 2. PMID 24189107
- [Background] Ibarra JM, Ge HY, Wang C, Martinez Vizcaino V, Graven-Nielsen T, Arendt-Nielsen L. Latent myofascial trigger points are associated with an increased antagonistic muscle activity during agonist muscle contraction. J Pain. 2011 Dec;12(12):1282-8. doi: 10.1016/j.jpain.2011.09.005. Epub 2011 Nov 11. PMID 22078789
- [Background] Baima J, Isaac Z. Clean versus sterile technique for common joint injections: a review from the physiatry perspective. Curr Rev Musculoskelet Med. 2008 Jun;1(2):88-91. doi: 10.1007/s12178-007-9011-2. PMID 19468878
- [Background] Administration FaD. Code of Federal Regulations Title 21. 2018; https://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfcfr/cfrsearch.cfm?fr=880.5580. Accessed March 24, 2019.